CLINICAL TRIAL: NCT01657435
Title: Ceramax™ Ceramic-on-Ceramic Acetabular Cup Prothesis System
Brief Title: 28mm Ceramic-on-Ceramic Total Hip Replacement Study
Acronym: COC28
Status: Terminated | Type: Observational
Why Stopped: Adequate data to satisfy PAS as agreed to with FDA 02OCT2019
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 09001
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Non-inflammatory Degenerative Joint Disease; Osteoarthritis; Avascular Necrosis; Post-traumatic Arthritis
Keywords: Total hip replacement; Total hip arthroplasty; Hip joint replacement; Hip prosthesis replacement
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ceramax COC 28mm Acetabular Cup: The 28 mm ceramic acetabular bearing insert component is manufactured from high purity, dense alumina matrix composite ceramic. The inserts secure to DePuy's Pinnacle acetabular shells by means of an interlocking mechanical taper. The Pinnacle acetabular shell is a hemispherical type acetabulum replacement prosthesis, is available in a range of outer diameter (OD) sizes, and is used with a 28mm femoral head. Pinnacle 100 shells will be used in this study. The BIOLOX® delta ceramic femoral head components are manufactured from the same ceramic material as the acetabular bearing insert components. The femoral head is secured to the femoral stem component with an interlocking taper.
  Interventions: Device: Ceramax Acetabular System

INTERVENTIONS:
Device: Ceramax Acetabular System — 28mm Ceramic-on-ceramic Acetabular Cup System
  Other Names: Ceramic-on-ceramic 28 mm Acetabular Cup

SUMMARY:
This study is intended to gather medium (0-5 years) and long-term (6-10 years) information regarding the performance and safety of the commercially available Ceramax™ Ceramic on Ceramic Total Hip System. This is a two-phased study consisting of a clinical follow-up phase and a clinical outcomes phase.

In Phase One (0-5 years), diagnostic, demographic and operative information will be gathered for each subject enrolled in this study. In addition, Harris Hip Evaluations, subjective evaluations and radiographs will be completed annually.

In Phase Two (6 - 10 years), a subjective outcomes questionnaire and a SF-12 Health Survey will be mailed to subjects annually.

DETAILED DESCRIPTION:
This is a prospective, non-randomized study of the 28mm Ceramic on Ceramic (COC) device. This study will follow each subject through 10 years postoperatively and will consist of:

1. a clinical follow-up phase and
2. a clinical outcomes phase.

Radiographic and clinical follow-up exams will take place at six-weeks, six-months and then annually through year 5 for each subject. For years 6 - 10, a communication will be sent to each subject in order to collect survivorship and general health information. This communication will ask whether the COC device is still in vivo and, if not, when the revision surgery took place, why, and which components were removed, if applicable. In addition, subjects will be asked to complete a SF-12 Health Survey at each 6 to 10-year follow-up interval. A self-addressed, stamped envelope will be provided to facilitate information return and privacy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were previously enrolled in the COC28 IDE study, or
* Newly recruited individuals who are qualified based on the approved labeling of the device, and;
* Individuals who are willing and able to provide informed patient consent for participation in the study;
* Individuals who are willing and able to return for follow-up as specified by the study protocol; and
* Individuals who are willing and able to complete the Hip Outcomes questionnaire and SF-12 Health Survey as specified by the study protocol

Exclusion Criteria:

* In the opinion of the Investigator, the individual does not qualify based upon approved labeling requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males and females who are appropriate candidates for primary hip replacement o any age, with non-inflammatory degenerative joint disease or: males and females that had a primary hip replacement with CERAMAX as part of the 28 mm IDE study.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Survivorship | 10 years
  The primary outcome measure is that the 10-year Kaplan-Meier survivorship estimate of the COC 28mm implanted hips will be a minimum of 90% (as recommended by National Institute of Clinical Excellence [NICE]). Based on an anticipated margin of error (ie. one-half the width of the confidence interval) of 7%, the lower 95% confidence interval will be no worse than 83%.

SECONDARY OUTCOMES:
Harris Hip Score | 5 years
  At five years, the Harris Hip Score must be > 80 points or higher and the Harris Hip pain assessment must be mild or no pain.
Radiographic | 5 years
  At 5 years, secondary radiographic outcome measures will include:
  * No radiolucencies >2mm in any zone in any post-operative interval;
  * No acetabular cup migration >4mm;
  * No change in cup inclination angle >4 degrees when compared to immediate post-operative angle; and
  * No osteolysis.
Survivorship | 5 years
  At 5 years, the secondary outcome measure will include no components removed for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Tammy L ODell, BS CCRC CCRA, Study Director — DePuy Orthopaedics
Locations (13):
- United States (12):
  - Joint Surgeons of Sacremento, Sacramento, California
  - Colorado Joint Replacement, Denver, Colorado
  - Fort Collins, Colorado
  - Florida University, Gainesville, Florida
  - FOI Florida Orthopaedic Institute, Tampa, Florida
  - New England Baptist Hospital, Boston, Massachusetts
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Duke University, Durham, North Carolina
  - OrthoCarolina, Winston-Salem, North Carolina
  - Cardinal Orthopaedic Institute, Columbus, Ohio
  - UPenn, Philadelphia, Pennsylvania
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia
- McGill University - Jewish General Hospital, Montreal, Quebec, Canada